CLINICAL TRIAL: NCT06244875
Title: Collection Biologique Des Atteintes Neurocognitives
Brief Title: Biological Collection of Neurocognitive Disorders
Acronym: BioCogBank
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230999
Record Dates: First submitted 2023-12-12; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-12

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients followed in the memory clinic
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Blood and cerebrospinal fluid sampling during the diagnostic visit

SUMMARY:
The development of biological biomarkers reflecting neuropathology has enhanced the diagnostic precision of Alzheimer's disease over the past decade, compared to the clinical diagnosis that suffers from low specificity. Patients undergoing evaluation in specialized memory clinics suspected of major or minor neurocognitive disorder are notably examined through a lumbar puncture to measure beta-amyloid 42, beta-amyloid 40, total tau, and phosphorylated tau in the cerebrospinal fluid (CSF). The purpose of this clinico-biological collection is to better characterize the existing biomarkers used in clinical practice, as well as the development of new diagnostic or prognostic biomarkers for neurodegenerative diseases causing neurocognitive disorder (Alzheimer's disease, Lewy body disease, frontotemporal lobar degeneration, in particular).

The primary objective is to gain a better understanding of conventional biomarkers and to develop new diagnostic and prognostic biomarkers for neurocognitive diseases: establishing a prospective clinico-biological collection of patients evaluated in clinical practice for a neurocognitive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Not under legal guardianship
* Clinical indication for blood and cerebrospinal fluid (CSF) biomarkers measurement during a day hospital stay for Alzheimer's disease (beta-amyloid peptide, tau protein).
* Signature of the research consent form.

Exclusion Criteria:

* Not affiliated with a social security scheme.
* Patient under State Medical Aid (AME).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in the memory clinic at the Center for Cognitive Neurology of Lariboisière Hospital (APHP) or at the memory clinic of Bretonneau Hospital (APHP), with a clinical indication for the measurement of blood and cerebrospinal fluid (CSF) biomarkers (day hospital for the diagnosis of a neurocognitive disorder).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2044-02-01 (Estimated); Study Completion 2044-02-01 (Estimated)

PRIMARY OUTCOMES:
Identification of new biomarkers for neurodegenerative diseases | Up to 10 years

SECONDARY OUTCOMES:
Description of the level of usual biomarkers by type of dementia | Up to 10 years
Evaluation of the relationship between biomarker levels and cognitive evolution measured in routine care | Up to 10 years
Comparison of biomarker levels in neurodegenerative pathologies and psychiatric pathologies with cognitive expression | Up to 10 years

IPD SHARING:
Plan to Share IPD: Undecided